CLINICAL TRIAL: NCT05726721
Title: Profiling the Dynamic of Binge Eating Disorder (BED): a Longitudinal Study Examining the Influence of Emotion Regulation, Executive Function, Eating Pattern on BED and Outcome (PRODY-BED)
Brief Title: Profiling the Dynamic of Binge Eating Disorder (PRODY-BED)
Acronym: PRODY-BED
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Kompetencecenter for Spiseforstyrrelser (Unknown)
Responsible Party: Principal Investigator, Loa Clausen, Senior Researcher, Aarhus University Hospital
Other Study IDs: PRODY-BED
Record Dates: First submitted 2022-12-15; First posted 2023-02-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Binge-Eating Disorder; Emotion Regulation; Executive Dysfunction; Eating Behavior; Depressive Symptoms
Keywords: psychotherapy; Adults; binge eating disorder; emotion regulation; executive function
MeSH Terms: conditions — Binge-Eating Disorder; Emotional Regulation; Feeding Behavior; Depression | interventions — Therapeutics; Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Treatment as usual, Psychotherapy — The three treament sites will offer psychotherapy as usual. All including elements of cognitive behavioral therapy and some sites also additional elements from either narrative therapy or interpersonal therapy

SUMMARY:
The goal of this observational study is to explore if different and specific profiles can be identified in adults with binge eating disorder (BED) depending on their additional eating pathology, emotion regulation and executive functions. The main questions it aims to answer are:

* Is there different and specific subgroups of patients with BED according to baseline profiles in emotion regulation, executive function and additional eating pathology (including restriction, chaotic eating, grazing and eating on external cues)?
* Are subgroups of individuals with BED (based on identified profiles) associated with outcome at end of treatment and follow-up?
* What is the trajectories in remission rates of specific symptom dimensions (eating disorder pathology, emotion regulation, executive function, and depressive symptoms) in individuals with BED and is there specific trajectory profiles in these dimensions?
* Is early changes in specific symptom dimensions (eating pathology, emotion regulation, executive function, or depression) associated with outcome of BED? Participants will be asked to fill in questionnaires before treatment as usual, 10 weeks into treatment, at end of treatment and at 6- and 12-month follow-up.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is a severe eating disorder characterized by recurrent episodes of binge eating, where control over eating is lost and huge amounts of food are eaten within a short period of time. Hence, weight issues are often inevitable and overweight is common, as are social, mental as well as physical problems.

The etiology of binge eating disorder is an interplay of neurobiological and environmental factors. Overall pathological eating, including grazing, external, emotional or restrictive eating, is associated with binge eating, and so is dysregulation in the reward center, impairment of executive functions and emotion regulation. The investigators suggest that it is possible to identify specific profiles driving binge eating, depending on the severity of these dimensions, and that these profiles might predict the outcome of treatment. The investigators also suggest that early change in general eating pattern, emotion regulation, and depressive symptoms is associated with binge eating outcome. These assumptions will be tested in a sample of adults in treatment for BED at one of three sites using questionnaires before, during and after treatment, incl. 6- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+,
* diagnosed with Binge eating Disorder,
* and offered treatment at on of the inclusion sites.

Exclusion Criteria:

* Severe psychiatric comorbidity (e.g. psychosis, severe developmental disorder, severe cogntive impairement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18+ years diagnosed with BED, accepted for treatment at one of the three sites, and accepting participation.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Subgroups of BED-profiles | Baseline data
  Subgroups of BED-profiles depending on degree and type of additional eating pathology measured by DEBQ (Dutch Eating Behaviour Questionnaire), emotion regulation problems measured by DERS-16 (Difficulties in Emotion Regulation Scale), and executive problems mesured by BRIEF-A .
Binge eating episodes EoT | At end of therapy up to 30 weeks
  Number of binge eating episodes
Binge eating episodes FU6m | At 6-month follow-up
  Number of binge eating episodes
Binge eating episodes FU12m | At 12-month follow-up
  Number of binge eating episodes

SECONDARY OUTCOMES:
Eating disorder pathology | At end of treatment up to 30 weeks
  Overall self-reported eating disorder pathology measured by the total score of Eating Disoder Examination Questionnaire (EDE-Q), minimum score 0, maximum score 6, higher scores indicating eating pathology
Eating disorder pathology | At 6-month follow-up
  Overall self-reported eating disorder pathology measured by the total score of EDE-Q, minimum score 0, maximum score 6, higher scores indicating eating pathology
Eating disorder pathology | At 12-month follow-up
  Overall self-reported eating disorder pathology measured by the total score of EDE-Q, minimum score 0, maximum score 6, higher scores indicating eating pathology
Functional impairment | At end of treatment up to 30 weeks
  Self-reported functional impairment measured by the total score of WSAS, minimum score 0, maximum score 8, higher scores indicating more impairment
Functional impairment | At 6-month follow-up
  Self-reported functional impairment measured by the total score of WSAS, minimum score 0, maximum score 8, higher scores indicating more impairment
Functional impairment | At 12-month follow-up
  Self-reported functional impairment measured by the total scorer of WSAS, minimum score 0, maximum score 8, higher scores indicating more impairment
Well-being | At end of treatment up to 30 weeks
  Self-reported well-being measured by the total score of WHO-5, minimum score 0, maximum score 25, with lower scores indicating worst imaginable well-bing
Well-being | At 6-month follow-up
  Self-reported well-being measured by the total score of WHO-5, minimum score 0, maximum score 25, with lower scores indicating worst imaginable well-bing
Well-being | At 12-month follow-up
  Self-reported well-being measured by the total score of WHO-5, minimum score 0, maximum score 25, with lower scores indicating worst imaginable well-bing
Trajectories of binge eating | From baseline to 12-month follow-up
  Trajectories of frequency of binge eating across time measured by self-reported binge eating in Eating Disorder Examination questionnaire (EDE-Q)
Trajectories of restrictive eating | From baseline to 12-month follow-up
  Trajectories of restrictive eating across time measured by the DEBQ restraint eating scale, minum score 1, maximum score 5, higher scores indicating more restricted eating
Trajectories of emotional eating | From baseline to 12-month follow-up
  Trajectories of emotional eating across time measued by the DEBQ emotional eating scale, minimum score 1, maximum score 5, higher scores indicating more emotional eating
Trajectories of eating on external cues | From baseline to 12-month follow-up
  Trajectories of eating on external cues across time measured by the DEBQ external eating scale, minimum score 1, maximum score 5, higher scores indicating more eating on external cues
Trajectories of grazing | From baseline to 12-month follow-up
  Trajectories of grazing across time measured by the total score of the Grazing Questionnaire, minimum 0, maximum 28, higher scores indcating greater grazing behavior
Trajectories of emotional regulation | From baseline to 12-month follow-up
  Trajectories of emotional regulation across time measured by the total score of DERS-16, minimum score 16, maximum score 80, higher socres indicating greater diffuculties
Trajectories of executive function | From baseline to 12-month follow-up
  Trajectories of executive function across time measured by the BRIEF-A (Behavior rating inventory of Executive Function Adult version) Global Executive Composite T-Scores, minimum score 0, maximum score 90, higher scores indicating executive problems
Trajectories of depression | From baseline to 12-month follow-up
  Trajectories of depression across time measured by Beck Depression Inventory 2, minimum score 0, maximum score 63, higher scores indicating more depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Loa Clausen, PhD, Principal Investigator — Aarhus University Hospital, Psychiatry
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Psychiaty, Aarhus, Central Jutland
  - Aalborg University Hospital, Aalborg
  - Kompetencecenter, Copenhagen NV

IPD SHARING:
Plan to Share IPD: No
Due til Danish legislation individual participant data wil not be available to researchers outside the research group.